CLINICAL TRIAL: NCT07121296
Title: Screen, Treat and Retain People With Primary Meth Use Disorder at MMT Clinics
Acronym: STAR-OM+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Giang Le Minh, Dean of the Institute of Preventive Medicine and Public Health, Hanoi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3R01DA050486-05S1 (NIH); 3R01DA050486-05S1 (NIH)
Record Dates: First submitted 2025-07-22; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Methamphetamine Use Disorder
Keywords: methamphetamine; methadone; Vietnam; STAR-OM

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Contingency management for Substance use (Experimental): Participants receive contingency management for their abstinence over 12 weeks
  Interventions: Behavioral: Contingency management for substance use
- Group-based Matrix plus contingency management (Experimental): Participants receive group-based Matrix counseling and contingency management for their attendance in group counseling sessions
  Interventions: Behavioral: Contingency management for attendance; Behavioral: Group-based Matrix counseling
- Individual-based Matrix plus contingency management (Experimental): Participants receive individual-based Matrix counseling and contingency management for their attendance in individual counseling sessions
  Interventions: Behavioral: Contingency management for attendance; Behavioral: Individual-based Matrix counseling

INTERVENTIONS:
Behavioral: Contingency management for substance use — Participants receive escalating incentives for each consecutive negative weekly urine drug screen.
  Arms: Contingency management for Substance use
Behavioral: Contingency management for attendance — Participants receive escalating incentives for each consecutive counseling session they attended.
  Arms: Group-based Matrix plus contingency management; Individual-based Matrix plus contingency management
Behavioral: Group-based Matrix counseling — Group-based Matrix counseling
  Arms: Group-based Matrix plus contingency management
Behavioral: Individual-based Matrix counseling — Individual-based Matrix counseling
  Arms: Individual-based Matrix plus contingency management

SUMMARY:
This study is built upon the STAR-OM study (R01 DA050486) to assess if providing psycho-behavioral interventions and medications for people with primary methamphetamine use disorder (MUD) and without opioid use disorder (OUD) at methadone clinics is feasible and acceptable. In Vietnam and many U.S. settings, clinics providing medication for OUD (especially methadone clinics) are the only viable option for evidence-based addiction treatment. Importantly, many of these clinics are at primary care level and therefore accessible to people with primary MUD, who are in dire need for effective treatment. Furthermore, providers in methadone clinics are capable of conducting psycho-behavioral interventions, which remain the first line of treatment for MUD, and prescribing medications should these medications become available and approved by authorities. It remains unknown, however, if methadone clinics could serve as treatment facilities for those with primary MUD. This Supplement to the STAR-OM study will 1) assess the feasibility and acceptability of three recruitment strategies to enroll people with MUD and without OUD in MUD treatment at methadone clinics and 2) explore the feasibility and acceptability of providing psycho-behavioral interventions as well as challenges in providing medications at methadone clinics for people with MUD and without OUD. In Aim 1, the study will screen 600 people with primary MUD recruited through three strategies (peer outreach, snowballing and social media) over 3 months to enroll 60 people with MUD and without OUD into the study interventions. Participants will be screened at MMT clinics for meth use and readiness for MUD intervention. The study team will monitor recruitment rate for each strategy to assess feasibility. Acceptability will be assessed through focus group discussions with people who support recruitment (N=2 focus group with 12-16 participants), in-depth interviews with individuals eligible for enrollment and agree or decline to participate in the study interventions (N=15, 5 per recruitment strategy). In Aim 2, consenting participants will be randomized 1:1:1 into three arms of interventions over 12 weeks: (1) contingency management only; (2) group-based Matrix plus contingency management; and (3) individual-based Matrix plus contingency management. All participants will be required to provide urine samples randomly once a week. The investigators will monitor participation and retention rate in each treatment arm and completion of urine drug screens to assess feasibility. Acceptability will be assessed through post-intervention in-depth interviews with 15 participants, focus groups with methadone providers who deliver behavioral interventions (N = 1 focus group with 6-8 participants), and in-depth interviews with policy makers at national and city levels (N=5). In addition, participants will be asked in these interviews and focus groups about the challenges and facilitators of providing medications for treatment of MUD at MMT clinics should they become available. Findings from this Supplement will be used to prepare for a larger trial to assess effectiveness of implementing psycho-behavioral interventions for people with primary MUD and without OUD at methadone clinics.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18
* ASSIST ≥ 10 OR urine drug screen positive with meth
* Urine drug screen negative with opioid and methadone
* Willing to participate in study interventions at selected MMT clinics

Exclusion Criteria:

* Unable to read and write Vietnamese
* Being incapable of understanding questions and research processes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates for screening and for enrollment to measure feasiblity of recruitment | Over the 3-month recruitment period
  Feasibility will be evaluated 1) by recruitment rate for screening at selected methadone clinics and 2) by recruitment rate for the study interventions among those screened. Feasibility is defined as at least 50% of those approached agree to participate in screening and among those eligible at least 50% agree to participate in the study interventions.
Themes of perceptions regarding each recruitment strategy from focus groups and in-depth interviews to assess the acceptability of recruitment strategies | Two weeks at the end of the 3-month recruitment period
  Acceptability will be assessed by perceived challenges and facilitators of recruitment and enrollment. Two focus group discussions will be organized with 12-16 participants who support recruitment and 15 in-depth interviews (5 per recruitment strategy) will be conducted with individuals eligible for enrollment and agree or decline to participate in the study interventions. Themes of positive perceptions of recruitment and enrollment are considered indicators of acceptability.
Rate of attendance in intervention sessions, rate of retention and rate of completion of urine drug screen to measure the feasibility of providing interventions at methadone clinics | Up to 12 weeks per participants from enrollment to completion of intervention
  Feasibility is defined by the rate of attendance in intervention sessions, retention in treatment and completion of urine drug screens (UDS). The STAR-OM data indicated that in any given week, approximately 85% of participants attended Matrix sessions and 88% completed UDS visits. Acknowledging the challenges facing people with primary MUD and without OUD in attending intervention sessions at methadone clinics regularly over 12 weeks, the study intervention is deemed feasible if the study reaches 70% of overall intervention attendance and 70% of overall UDS completion.
Themes of perceptions from focus groups and in-depth interviews regarding how acceptable it is to provide intervention at methadone clinics and percentage of participants indicating that the intervention is satisfactory | Upon the completion of intervention (Week 12) per selected participants
  Acceptability is defined as a common theme of positive perceptions among both participants and providers of providing each type of intervention, behavioral or medication, for people with primary MUD but without OUD at methadone clinics. Acceptability will be assessed through post-intervention in-depth interviews with 15 participants, focus groups with methadone providers who deliver behavioral interventions (N = 1 focus group with 6-8 participants), and in-depth interviews with policy makers at national and city levels (N=5). Acceptability is also defined by 70% of participants indicating that the intervention is agreeable or satisfactory in the 12-week assessment.

SECONDARY OUTCOMES:
Number of meth use days, cost for meth use in the past 30 days and urine test results over 12 weeks of intervention | From baseline to 12-week follow-up
  Changes in reported meth use and urine drug screen results between baseline and 12-week follow-up. The study team uses Timeline Follow-back method to collect data on the number of meth use days and the cost for meth use in the past 30 days at baseline and at 12-week follow-up visit. Participants undergo one weekly urine drug screen throughout the 12 weeks of intervention.
Depression, Anxiety and Stress Scale version with 21 items (DASS-21) | From baseline to 12-week follow-up
  Changes in the mean scores of each of the subscales in the Depression, Anxiety and Stress Scale version with 21 items (DASS-21) between baseline and 12-month follow-up. DASS-21 has 3 subscales for depression, anxiety and stress. Each subscale has 7 items, rated on a 4-point Likert scale. Scores (after multiplying by 2) range from 0 to 42. Lower scores mean better mental health status.
Rapid HIV testing | From baseline to 12-week follow-up
  Changes in HIV status as determined by rapid HIV testing between baseline and 12-week follow-up
Chesney (1997)'s questionnaire on HIV sexual risk behaviors related to substance use | From baseline to 12-week follow-up
  HIV sexual risk behaviors related to substance use are measured using Chesney et al. (1997)'s questionnaire. Injection practices in relation to meth use are also inquired. This section consists of 8 questions asking about unprotected sexual behaviors and injection equipment sharing. The unit of measure is percentage of participants indicating yes for each risk behavior.
Themes of perceptions from focus groups and in-depth interviews regarding how feasible it is to provide medications to treat methamphetamine use disorder | Within 2 weeks after the last participant completes the intervention
  Feasibility of providing medications at methadone clinics for people with primary methamphetamine use disorder and without opioid use disorder is assessed qualitatively and defined as a common theme of positive perceptions among MMT providers and policy makers (1 focus group with 6-8 MMT providers, and 5 in-depth interviews with policy makers at national and city levels).
Themes of perceptions from focus groups and in-depth interviews regarding how acceptable it is to provide medications to treat methamphetamine use disorder | Within 2 weeks after the last participant completes the intervention
  Acceptability of providing medications at methadone clinics for people with primary methamphetamine use disorder and without opioid use disorder is assessed qualitatively and defined as a common theme of positive perceptions among MMT providers and policy makers (1 focus group with 6-8 MMT providers, and 5 in-depth interviews with policy makers at national and city levels).

CONTACTS AND LOCATIONS:
Overall Officials: Giang M. Le, MD, PhD, Principal Investigator — Hanoi Medical University
Locations (1):
- Hanoi Medical University, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Des Jarlais DC, Arasteh K, Huong DT, Oanh KTH, Feelemyer JP, Khue PM, Giang HT, Thanh NTT, Vinh VH, Le SM, Vallo R, Quillet C, Rapoud D, Michel L, Laureillard D, Moles JP, Nagot N; DRIVE Study Team. Using large-scale respondent driven sampling to monitor the end of an HIV epidemic among persons who inject drugs in Hai Phong, Viet Nam. PLoS One. 2021 Nov 18;16(11):e0259983. doi: 10.1371/journal.pone.0259983. eCollection 2021. PMID 34793523
- [Background] Giang HT, Duc NQ, Khue PM, Quillet C, Oanh KTH, Thanh NTT, Vallo R, Feelemyer J, Vinh VH, Rapoud D, Michel L, Laureillard D, Moles JP, Jarlais DD, Nagot N, Huong DT. Gender Differences in HIV, HCV risk and Prevention Needs Among People who Inject drug in Vietnam. AIDS Behav. 2023 Jun;27(6):1989-1997. doi: 10.1007/s10461-022-03932-x. Epub 2022 Nov 28. PMID 36441408
- [Background] Bolivar HA, Klemperer EM, Coleman SRM, DeSarno M, Skelly JM, Higgins ST. Contingency Management for Patients Receiving Medication for Opioid Use Disorder: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2021 Oct 1;78(10):1092-1102. doi: 10.1001/jamapsychiatry.2021.1969. PMID 34347030
- [Background] Weinstock J, Alessi SM, Petry NM. Regardless of psychiatric severity the addition of contingency management to standard treatment improves retention and drug use outcomes. Drug Alcohol Depend. 2007 Mar 16;87(2-3):288-96. doi: 10.1016/j.drugalcdep.2006.08.027. Epub 2006 Sep 26. PMID 17005329
- [Background] Miguel AQ, Madruga CS, Cogo-Moreira H, Yamauchi R, Simoes V, da Silva CJ, McPherson S, Roll JM, Laranjeira RR. Contingency management is effective in promoting abstinence and retention in treatment among crack cocaine users in Brazil: A randomized controlled trial. Psychol Addict Behav. 2016 Aug;30(5):536-543. doi: 10.1037/adb0000192. Epub 2016 Jul 21. PMID 27442691
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Chesney MA, Chambers DB, Kahn JO. Risk behavior for HIV infection in participants in preventive HIV vaccine trials: a cautionary note. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Dec 1;16(4):266-71. doi: 10.1097/00042560-199712010-00007. PMID 9402073
- [Background] Twitchell GR, Huber A, Reback CJ, Shoptaw S. Comparison of General and Detailed HIV Risk Assessments Among Methamphetamine Abusers. AIDS Behav. 2002;6(2):153-162. doi:10.1023/A:1015449231848
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Le MTH, Tran TD, Holton S, Nguyen HT, Wolfe R, Fisher J. Reliability, convergent validity and factor structure of the DASS-21 in a sample of Vietnamese adolescents. PLoS One. 2017 Jul 19;12(7):e0180557. doi: 10.1371/journal.pone.0180557. eCollection 2017. PMID 28723909
- [Background] McGregor C, Srisurapanont M, Mitchell A, Longo MC, Cahill S, White JM. Psychometric evaluation of the Amphetamine Cessation Symptom Assessment. J Subst Abuse Treat. 2008 Jun;34(4):443-9. doi: 10.1016/j.jsat.2007.05.007. Epub 2007 Jul 13. PMID 17629443
- [Background] Sobell LC, Sobell MB. Timeline follow-back: A technique for assessing self-reported alcohol consumption. In: Measuring Alcohol Consumption: Psychosocial and Biochemical Methods. Totowa, NJ, US: Humana Press/Springer Nature; 1992:41-72. doi:10.1007/978-1-4612-0357-5_3
- [Background] Giang LM, Li MJ, Okafor CN, Diep NB, Shoptaw SJ. Correlates of methamphetamine use severity among patients receiving methadone maintenance treatment for opioid use disorder in Vietnam. J Subst Abuse Treat. 2022 Jan;132:108461. doi: 10.1016/j.jsat.2021.108461. Epub 2021 May 7. PMID 34098204
- [Background] Hoang TA. Civil society organisations' roles in health development in Vietnam: HIV as a case study. Glob Public Health. 2013;8 Suppl 1:S92-103. doi: 10.1080/17441692.2013.811530. Epub 2013 Jul 4. PMID 23822631
- [Background] Nguyen Bich D, Korthuis PT, Nguyen Thu T, Van Dinh H, Le Minh G. HIV Patients' Preference for Integrated Models of Addiction and HIV Treatment in Vietnam. J Subst Abuse Treat. 2016 Oct;69:57-63. doi: 10.1016/j.jsat.2016.07.003. Epub 2016 Jul 19. PMID 27568511
- [Background] Des Jarlais DC, Feelemyer J, Arasteh K, Huong DT, Oanh KTH, Khue PM, Giang HT, Thanh NTT, Moles JP, Vinh VH, Vallo R, Quillet C, Rapoud D, Michel L, Laureillard D, Nagot N; DRIVE Study Team. The methamphetamine epidemic among persons who inject heroin in Hai Phong, Vietnam. J Subst Abuse Treat. 2021 Jul;126:108320. doi: 10.1016/j.jsat.2021.108320. Epub 2021 Feb 4. PMID 34116818
- [Background] Giang LM, Trang NT, Thuy DT, Nguyen HH, Diep NB, Van HTH, Truc TT, Reback CJ, Li M, Van Dung D, Shoptaw S. Using ADAPT-ITT framework to tailor evidence-based interventions for addressing methamphetamine use among methadone patients in Vietnam. Drug Alcohol Rev. 2023 Nov;42(7):1667-1679. doi: 10.1111/dar.13739. Epub 2023 Aug 23. PMID 37614129
- [Background] Tran BX, Nguyen QL, Nguyen LH, Phan HTT, Le HT, Tran TD, Vu TTM, Latkin CA. Expanding co-payment for methadone maintenance services in Vietnam: the importance of addressing health and socioeconomic inequalities. BMC Health Serv Res. 2017 Jul 12;17(1):480. doi: 10.1186/s12913-017-2405-y. PMID 28701208
- [Background] Farhoudian A, Razaghi E, Hooshyari Z, Noroozi A, Pilevari A, Mokri A, Mohammadi MR, Malekinejad M. Barriers and Facilitators to Substance Use Disorder Treatment: An Overview of Systematic Reviews. Subst Abuse. 2022 Aug 29;16:11782218221118462. doi: 10.1177/11782218221118462. eCollection 2022. PMID 36062252
- [Background] Ginley MK, Pfund RA, Rash CJ, Zajac K. Long-term efficacy of contingency management treatment based on objective indicators of abstinence from illicit substance use up to 1 year following treatment: A meta-analysis. J Consult Clin Psychol. 2021 Jan;89(1):58-71. doi: 10.1037/ccp0000552. PMID 33507776
- [Background] Moszczynska A. Current and Emerging Treatments for Methamphetamine Use Disorder. Curr Neuropharmacol. 2021;19(12):2077-2091. doi: 10.2174/1570159X19666210803091637. PMID 34344291
- [Background] Han B, Compton WM, Jones CM, Einstein EB, Volkow ND. Methamphetamine Use, Methamphetamine Use Disorder, and Associated Overdose Deaths Among US Adults. JAMA Psychiatry. 2021 Dec 1;78(12):1329-1342. doi: 10.1001/jamapsychiatry.2021.2588. PMID 34550301
- [Background] Naji L, Dennis B, Rosic T, Wiercioch W, Paul J, Worster A, Thabane L, Samaan Z. Mirtazapine for the treatment of amphetamine and methamphetamine use disorder: A systematic review and meta-analysis. Drug Alcohol Depend. 2022 Mar 1;232:109295. doi: 10.1016/j.drugalcdep.2022.109295. Epub 2022 Jan 11. PMID 35066460
- [Background] Colfax GN, Santos GM, Das M, Santos DM, Matheson T, Gasper J, Shoptaw S, Vittinghoff E. Mirtazapine to reduce methamphetamine use: a randomized controlled trial. Arch Gen Psychiatry. 2011 Nov;68(11):1168-75. doi: 10.1001/archgenpsychiatry.2011.124. PMID 22065532
- [Background] Bakouni H, Sharafi H, Bahremand A, Drouin S, Ziegler D, Bach P, Le Foll B, Schutz CG, Tardelli V, Ezard N, Siefried K, Jutras-Aswad D. Bupropion for treatment of amphetamine-type stimulant use disorder: A systematic review and meta-analysis of placebo-controlled randomized clinical trials. Drug Alcohol Depend. 2023 Dec 1;253:111018. doi: 10.1016/j.drugalcdep.2023.111018. Epub 2023 Nov 4. PMID 37979478
- [Background] Coffin PO, Santos GM, Hern J, Vittinghoff E, Walker JE, Matheson T, Santos D, Colfax G, Batki SL. Effects of Mirtazapine for Methamphetamine Use Disorder Among Cisgender Men and Transgender Women Who Have Sex With Men: A Placebo-Controlled Randomized Clinical Trial. JAMA Psychiatry. 2020 Mar 1;77(3):246-255. doi: 10.1001/jamapsychiatry.2019.3655. PMID 31825466
- [Background] Knight R, Karamouzian M, Carson A, Edward J, Carrieri P, Shoveller J, Fairbairn N, Wood E, Fast D. Interventions to address substance use and sexual risk among gay, bisexual and other men who have sex with men who use methamphetamine: A systematic review. Drug Alcohol Depend. 2019 Jan 1;194:410-429. doi: 10.1016/j.drugalcdep.2018.09.023. Epub 2018 Nov 3. PMID 30502543
- [Background] AshaRani PV, Hombali A, Seow E, Ong WJ, Tan JH, Subramaniam M. Non-pharmacological interventions for methamphetamine use disorder: a systematic review. Drug Alcohol Depend. 2020 Jul 1;212:108060. doi: 10.1016/j.drugalcdep.2020.108060. Epub 2020 May 13. PMID 32445927
- [Background] Trivedi MH, Walker R, Ling W, Dela Cruz A, Sharma G, Carmody T, Ghitza UE, Wahle A, Kim M, Shores-Wilson K, Sparenborg S, Coffin P, Schmitz J, Wiest K, Bart G, Sonne SC, Wakhlu S, Rush AJ, Nunes EV, Shoptaw S. Bupropion and Naltrexone in Methamphetamine Use Disorder. N Engl J Med. 2021 Jan 14;384(2):140-153. doi: 10.1056/NEJMoa2020214. PMID 33497547
- [Background] Giang LM, Trang NT, Diep NB, Thuy DTD, Thuy DT, Hoe HD, Van HTH, Truc TT, Nguyen HH, Lai NL, Linh PTD, Vi VTT, Reback CJ, Leibowitz A, Li L, Lin C, Li M, Do Van Dung, Shoptaw S. An adaptive design to screen, treat, and retain people with opioid use disorders who use methamphetamine in methadone clinics (STAR-OM): study protocol of a clinical trial. Trials. 2022 Apr 23;23(1):342. doi: 10.1186/s13063-022-06278-w. PMID 35461300